CLINICAL TRIAL: NCT02366806
Title: Impact of Individualized Radiotherapy Plan Review in Patients Receiving Adjuvant Radiotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 587842; CCRO035 (Other: UC Davis)
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; AJCC Stage 1, 2, 3; Educational Design; Radiation Therapy Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In-Depth Education: A. Standard radiotherapy discussion including rationale, number of fractions, side effects, +/- beam arrangements, potential and likely short and long-term toxicity, status checks, skin care, nursing and physician accessibility B. Radiotherapy plan review to include, but not limited to: beam arrangement, total dose, dose per fraction, target area(s), description of isodose lines, DVH review and discussion of prescription constraints for OARs

SUMMARY:
This study is being conducted to investigate the effect of a more in-depth education plan for patients with breast cancer. Patients will be randomized to receive either the standard education plan during their breast cancer treatment or they will receive in-depth education about their breast cancer treatment. In order to see what kind of effect the different education plans have, patients will fill out three identical questionnaires during the course of treatment.

DETAILED DESCRIPTION:
This study will be a prospective study of women receiving adjuvant radiation therapy for management of breast cancer at the University of California Davis. All patients will be staged according to the American Joint Committee on Cancer Seventh edition. Primary disease treatment information including surgical approach and utilization of adjuvant chemotherapy will be evaluated.

All patients will have a validated quality of life assessment (FACIT-TS-PS) completed at three time points during their radiation therapy process. The patients will be randomized at the time of completion of radiation plan approval by the treating radiation oncologist in a one to one fashion to either proceed with standard education or more extensive plan review. The radiation oncology quality assurance (QA) process will be blinded to the randomization of the patient.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of invasive breast cancer
2. AJCC stage 1, 2, 3 breast carcinoma
3. Patient deemed clinically appropriate for adjuvant breast or chest wall radiation following surgery
4. Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during radiation therapy
5. Patient must provide study specific informed consent prior to study entry
6. Breast implants allowed

Exclusion Criteria

1. Stage 4 breast cancer
2. Ductal carcinoma in situ
3. Patients treated with radiation for palliative intent
4. Prior treatment with radiation therapy to the ipsilateral breast or chest wall
5. Prior invasive non-breast malignancy (except non-melanomatous skin cancer, carcinoma in situ of the cervix) unless disease free for a minimum of 5 years prior to study entry
6. Prior invasive or in-situ carcinoma of the breast (-prior LCIS is eligible)
7. Diagnosis of DCIS

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is for women with breast cancer. All patients will be staged according to the American Joint Committee on Cancer Seventh edition. Primary disease treatment information including surgical approach and utilization of adjuvant chemotherapy will be evaluated.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Satisfaction measure | 3 months
  Questions on the survey will be analyzed to see if patients are more satisfied with the in-depth education compared to the standard education.

SECONDARY OUTCOMES:
Time measure | 3 Months
  The amount of time in the clinic office will be analyzed for the in-depth education plan as compared to the standard education plan.
Change in satisfaction over time | 3 months
  Questions on the survey will be analyzed from baseline to the end of treatment to see if there are differences over time between the in-depth education group and the standard education group.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States